CLINICAL TRIAL: NCT02895464
Title: Preoperative Home-based Exercise in Older People Before Colorectal Surgery - a Feasibility Study
Brief Title: Feasibility of Home-based Preoperative Exercise in Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm South General Hospital (Other)
Responsible Party: Principal Investigator, Elisabeth Rydwik, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LS1311-1462
Record Dates: First submitted 2016-08-09; First posted 2016-09-09 (Estimated); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The sessions will be led by a physiotherapist, in the older person's home. The sessions will consist of inspiratory muscle training with a resistance starting from 50% of their maximal capacity (30 breathes, 2 times/day). The training session will also consist of high-intensity individually adjusted functional strength and endurance training: chair-stand; stair climb/step up with weight belts, interval walking indoor and/or outdoor. This will be combined with functional task-exercises. The training will be conducted 2-3 times week, for at least two weeks or until they undergo surgery. During the remaining days, the participants will be instructed to follow the recommendation of 30 minutes of moderate physical activity per day, as well as to perform inspiratory muscle training.
  Interventions: Other: Exercise
- Control group (Other): The participants will receive ordinary preoperative information, but will also be encouraged to follow the recommendation of 150 minutes/week of moderate physical activity.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The sessions will be led by a physiotherapist, in the older person's home. The sessions will consist of inspiratory muscle training with a resistance starting from 50% of their maximal capacity (30 breathes, 2 times/day). The training session will also consist of high-intensity individually adjusted functional strength and endurance training: chair-stand; stair climb/step up with weight belts, interval walking indoor and/or outdoor. This will be combined with functional task-exercises. The training will be conducted 2-3 times week, for at least two weeks or until they undergo surgery. During the remaining days, the participants will be instructed to follow the recommendation of 30 minutes of moderate physical activity per day, as well as to perform inspiratory muscle training.

SUMMARY:
The purpose of the study is to evaluate the feasibility of recruitment procedure, intervention including compliance and the collaboration between in- and out patient clinics of preoperative home-based exercise in older people before colorectal surgery.

DETAILED DESCRIPTION:
The feasibility study will be conducted in order to evaluate the study design of a future RCT. Feasibility data will eg. consist of study flow description, number of eligible participants, included participants, patients and instructors satisfaction with the intervention, training compliance, reasons for drop-outs, and adverse events.

Patients waiting for colorectal surgery will be recruited and included after informed consent. Physical and respiratory function will be assessed at the hospital before the intervention, the day before surgery and the day before discharge. Data on postoperative complications, length of stay and mortality will be collected during the hospital stay. At baseline and six months after surgery, the participants will receive three questionnaires about level of independence in daily living, physical activity and health related quality of life. The intervention will be performed in the older person's home and consists of a combination of high-intensity respiratory training and individually adjusted functional exercise. Both groups will receive physical activity advice and malnutrition will be screened to optimize their nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* Age above 70, understand and speaks the Swedish language. Surgery due to cancer

Exclusion Criteria:

* Health status that contradicts participation in the study such as unstable heart disease or severe orthopaedic conditions that prohibits training and severe systematic illness.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Rydwik, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Stockholm South General Hospital, Stockholm, Sweden

REFERENCES:
- [Result] Karlsson E, Farahnak P, Franzen E, Nygren-Bonnier M, Dronkers J, van Meeteren N, Rydwik E. Feasibility of preoperative supervised home-based exercise in older adults undergoing colorectal cancer surgery - A randomized controlled design. PLoS One. 2019 Jul 2;14(7):e0219158. doi: 10.1371/journal.pone.0219158. eCollection 2019. PMID 31265476
- See also: Feasibility of preoperative supervised homebased exercise in older adults undergoing colorectal cancer surgery - A randomized controlled design — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0219158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients scheduled for colorectal cancer surgery at Stockholm South General Hospital were informed about the study and asked to participate. The screening for inclusion was undertaken from September 2016 to June 2018 by a surgeon and nurse at the weekly colorectal cancer conferences (CRC).
Pre-assignment Details: There were 66 eligible participants. Of those 66, 43 declined to participate due to: they did not want to delay surgery (n=6), felt it was too much stress (n=12), additional hospital visit (n=10), already exercising (n=3), no reason given (n=10), and could not be reached (n=2).
Period: Baseline
Arm/Group | Exercise Group | Control Group
Started | 11 | 12
Completed | 10 | 11
Not Completed | 1 | 1
Period: Follow-up
Arm/Group | Exercise Group | Control Group
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Group | Control Group | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Customized [Median (Inter-Quartile Range); unit: years] | 83.5 [76 to 85] | 74 [73 to 76] | 76 [73 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 4 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 10 | 11 | 21
Type of surgery approach [Count of Participants; unit: Participants]
  Open | 3 | 3 | 6
  Laparoscopic | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rate
Description: The recruitment rate is calculated by the number of participants allocated to either the exercise group or control group from the total number of eligible participants (n=66).
Time Frame: Baseline
Population: The number of participants allocated to each group [exercise group (n=11), control group (n=12), overall study (n=23)] by the total number of eligible participants (n=66).
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study: Total for the exercise group and control group.
Arm/Group | Overall Study
Number analyzed (Participants) | 66
Participants
  Exercise | 11
  Control | 12

2. Primary Outcome: Exercise Compliance
Description: Compliance with the exercise intervention was defined as the number of sessions attended out of planned sessions and was registered in the exercise logs by the physiotherapists in primary care. Only participants randomized to the exercise group were evaluated for this assessment.
Time Frame: At the end of the intervention, after 2-4 weeks
Population: The number of planned sessions and attended sessions.
Measure: Count of Units; unit: Number of exercise sessions
Units Other Than Participants: Number of exercise sessions
Groups:
- Planned Exercise Sessions: The total number of planned sessions that were included in the exercise intervention.
- Attended Exercise Sessions: The total number of attended sessions in the exercise intervention.
Arm/Group | Planned Exercise Sessions | Attended Exercise Sessions
Number analyzed (Participants) | 10 | 10
Number analyzed (Number of exercise sessions) | 60 | 60
Number of exercise sessions | 60 | 58

3. Primary Outcome: Acceptability
Description: Patients and instructors satisfaction with the intervention measured with a survey. Instructors were not enrolled. Only participants randomized to the exercise group were evaluated for this assessment.
Time Frame: At the end of the intervention, after 2-4 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Patients: Satisfaction with participating in the exercise program.
- Instructors: Satisfaction with instructing the exercise program.
Arm/Group | Patients | Instructors
Number analyzed (Participants) | 10 | 6
Participants | 10 | 5

4. Primary Outcome: Adverse Events
Description: Musculoskeletal-related events, cardiovascular episodes, falls and health care use that occurred during the exercise intervention before (pre)-surgery. Adverse events are only reported for the intervention group since the control group were a treatment as usual (TAU) group.
Time Frame: During the intervention, after 1-4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Exercise Group
Number analyzed (Participants) | 10
Participants | 3

5. Secondary Outcome: Six-minute Walk
Description: Meters completed, effort estimated
Time Frame: Baseline, before surgery (after 2-4 weeks), before discharge app 4-10 days after surgery
Measure: Median (95% Confidence Interval); unit: meter
Groups:
- Exercise Group: Intervention group
- Control Group: Treatment as usual, advice on physical activity
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 10 | 11
meter | 15 [-29 to 46] | -4 [-16 to 20]

6. Secondary Outcome: Inspiratory Muscle Strength
Description: Inspiratory muscle strength measured with MicroRPM.
Time Frame: Baseline, before surgery (after 2-4 weeks), before discharge app 4-10 days after surgery
Measure: Median (95% Confidence Interval); unit: cm H2O
Groups:
- Control Gorup: Treatment as usual, advice on physical activity
Arm/Group | Exercise Group | Control Gorup
Number analyzed (Participants) | 10 | 10
cm H2O | 17 [7 to 25] | -2 [-6 to 4]

7. Secondary Outcome: Chair-stand 30-sec
Description: Number of stands during 30 sec.
Time Frame: Baseline, before surgery (after 2-4 weeks), before discharge app 4-10 days after surgery
Measure: Median (95% Confidence Interval); unit: Stands per 30 sec
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 10 | 11
Stands per 30 sec | 3.5 [0 to 4] | 1 [-0.3 to 3.3]

8. Secondary Outcome: Walking Speed
Description: Normal walking speed was measured over 10 meters.
Time Frame: Baseline, before surgery (after 2-4 weeks), before discharge app 4-10 days after surgery
Measure: Median (95% Confidence Interval); unit: m/s
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 10 | 11
m/s | 0.09 [0 to 0.3] | 0.09 [-0.002 to 0.13]

9. Secondary Outcome: Postoperative Complications
Description: Clavien-Dindo, number of participants with at least one postoperative complication.
Time Frame: Within the first 30 days of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 10 | 11
Participants | 6 | 2

10. Secondary Outcome: Length of Stay
Description: Number of days admitted to the hospital
Time Frame: At discharge, 2-4 weeks after baseline
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Exercise Group | Control Group
Number analyzed (Participants) | 10 | 11
Days | 5 [4 to 6] | 6 [4 to 7]

ADVERSE EVENTS:
Time Frame: Three weeks
Arm/Group | Exercise Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 3/10 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise Group (N=10) | Control Group (N=11)
Dizziness (Vascular disorders) | 1 (2) | 0
Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — Joint pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2016-08-26): https://cdn.clinicaltrials.gov/large-docs/64/NCT02895464/Prot_000.pdf